CLINICAL TRIAL: NCT05388006
Title: MC198B, Phase II Study of a Combination Therapy of Acalabrutinib, Venetoclax and Durvalumab in Patients With Richter Transformation From Chronic Lymphocytic Leukemia (CLL)
Brief Title: Acalabrutinib, Venetoclax and Durvalumab for the Treatment of Richter Transformation From Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC198B; NCI-2022-02068 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20-006487 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2022-05-19; First posted 2022-05-24 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Chronic Lymphocytic Leukemia; Richter Syndrome; Small Lymphocytic Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — acalabrutinib; durvalumab; Immunoglobulin G; Disulfides; venetoclax; Specimen Handling; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (acalabrutinib, durvalumab, venetoclax) (Experimental): Patients receive acalabrutinib PO BID on days 1-28, durvalumab IV over 1 hour on day 1, and venetoclax PO QD on days 1-28 of each cycle. Cycles repeat every 28 days for 12 cycles in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE: Patients receive acalabrutinib PO BID and venetoclax PO QD on days 1-90 of each cycle. Cycles repeat every 90 days for 4 cycles in the absence of disease progression or unacceptable toxicity.
  Patients also undergo blood sample collection, bone marrow aspiration and biopsy, and PET/CT or CT throughout the study.
  Interventions: Drug: Acalabrutinib; Biological: Durvalumab; Drug: Venetoclax; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Positron Emission Tomography (PET); Procedure: Computed Tomography

INTERVENTIONS:
Drug: Acalabrutinib — Given PO
  Other Names: ACP-196; Bruton Tyrosine Kinase Inhibitor ACP-196; Calquence
Biological: Durvalumab — Given IV
  Other Names: Imfinzi; Immunoglobulin G1, Anti-(Human Protein B7-H1) (Human Monoclonal MEDI4736 Heavy Chain), Disulfide with Human Monoclonal MEDI4736 Kappa-chain, Dimer; MEDI-4736; MEDI4736
Drug: Venetoclax — Given PO
  Other Names: ABT-0199; ABT-199; ABT199; GDC-0199; RG7601; Venclexta; Venclyxto
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy
  Other Names: Biopsy of Bone Marrow
Procedure: Positron Emission Tomography (PET) — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; Pet Scan; positron emission tomography scan; PT
Procedure: Computed Tomography — Undergo PET/CT or CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized Tomography (CT) scan; CT

SUMMARY:
This phase II trial tests whether acalabrutinib, venetoclax, and durvalumab work in treating patients with Richter transformation from chronic lymphocytic leukemia or small lymphocytic lymphoma. Richter transformation is a rare condition in which chronic lymphocytic leukemia or small lymphocytic lymphoma changes into a fast-growing type of lymphoma. Acalabrutinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Venetoclax is in a class of medications called B-cell lymphoma-2 (BCL-2) inhibitors. It may stop the growth of cancer cells by blocking Bcl-2, a protein needed for cancer cell survival. Immunotherapy with monoclonal antibodies, such as durvalumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving acalabrutinib, venetoclax, and durvalumab may help improve survival in patients with Richter transformation.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine the progression free survival (PFS) at 6 months of the combination therapy of acalabrutinib, venetoclax, and durvalumab in patients with Richter transformation from chronic lymphocytic leukemia (CLL).

SECONDARY OBJECTIVES:

I. Determine the safety of the combination therapy of acalabrutinib, venetoclax and durvalumab in patients with Richter transformation from CLL.

II. Evaluate the overall response rate (ORR), complete response (CR) rate, and partial response (PR) rate of the above combination therapy.

III. Overall survival, PFS, and treatment free survival of this above combination therapy.

CORRELATIVE RESEARCH OBJECTIVES:

I. Determine the biomarkers that predict clinical response of this above combination therapy.

II. Determine the immune profiles of patients while receiving this combination of therapy.

OUTLINE:

Patients receive acalabrutinib orally (PO) twice daily (BID) on days 1-28, durvalumab intravenously (IV) over 1 hour on day 1, and venetoclax PO once daily (QD) on days 1-28 of each cycle. Cycles repeat every 28 days for 12 cycles in the absence of disease progression or unacceptable toxicity.

MAINTENANCE: Patients receive acalabrutinib PO BID and venetoclax PO QD on days 1-90 of each cycle. Cycles repeat every 90 days for 4 cycles in the absence of disease progression or unacceptable toxicity.

Patients also undergo blood sample collection, bone marrow aspiration and biopsy, and positron emission tomography (PET)/computed tomography (CT) or CT throughout the study.

After completion of study treatment, patients are followed up at 30 days and then every 90 days until 5 years from study enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years willing to provide consent and follow-up
* Diagnosis of CLL according to the International Workshop on Chronic Lymphocytic Leukemia (IWCLL) 2018 criteria (Hallek et al., 2018) or small lymphocytic lymphoma (SLL) according to the World Health Organization (WHO) 2008 criteria (Harris, 1999). This includes previous documentation of:

  * Biopsy-proven SLL according to WHO 2008 criteria, or
  * Diagnosis of CLL according to IWCLL 2018 criteria as evidenced by all of the following:

    * Peripheral blood B cell count of >= 5 x 10^9/L consisting of small to moderate size lymphocytes (If there are enough evidence to document the prior diagnosis of CLL, it is not required to meet the criteria of peripheral blood B cell count more than 5 x 10^9/L )
    * Immunophenotyping consistent with CLL defined as:

      * The predominant population of lymphocytes share both B-cell antigens (CD19, CD20 [typically dim expression], or CD23) as well as CD5 in the absence of other pan-T-cell markers (CD3, CD2, etc.)
      * Clonality as evidenced by kappa or lambda light chain expression (typically dim immunoglobulin expression) or other genetic method (e.g. immunoglobulin heavy chain variable [IGHV] analysis)

        * NOTE: Splenomegaly, hepatomegaly, or lymphadenopathy are not required for the diagnosis of CLL
    * Before diagnosing CLL or SLL, mantle cell lymphoma must be excluded by demonstrating a negative fluorescence in situ hybridization (FISH) analysis for t(11;14)(IgH/CCND1) on peripheral blood or tissue biopsy or negative immunohistochemical stains for cyclin D1 on involved tissue biopsy
    * If prior CLL diagnosis was confirmed, or CLL diagnosis was confirmed on bone marrow examination or tissue biopsy, peripheral blood B cell count less than 5 x 10^9/L is allowed
* Biopsy proven Richter's transformation of the CLL

  * NOTE: Previously treated patients including CLL therapy can be enrolled. If Richter's transformation (RT) developed from prior untreated CLL and has not received any RT directed therapy, then patient is not eligible
* Richter patients with prior or concurrent CLL diagnosis and do not have other option for standard therapy per treating physician's discretion
* Measurable disease can be detected in positron emission tomography (PET) or computed tomography (CT) (>= 1 cm in diameter)
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0, 1, or 2
* Absolute neutrophil count >= 0.7 x 10^9/L unless marrow was involved by CLL or RT, then absolute neutrophil count (ANC) >= 0.3 x 10^9/L (=< 14 days prior to registration)
* Platelet count >= 40 x 10^9/L unless marrow was involved by CLL or RT, then platelet >= 30 x 10^9/L without transfusion =< 1 week prior to study registration (=< 14 days prior to registration)
* Hemoglobin (Hgb) >= 8 unless marrow was involved by CLL or RT, then Hgb >= 7 without transfusion =< 1 week prior to study registration (=< 14 days prior to registration)
* Total bilirubin =< 1.5 x upper limit of normal (ULN) unless due to confirmed Gilbert's disease (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with their physician (=< 14 days prior to registration)

  * Note: If total bilirubin is > 1.5 x ULN, a direct bilirubin should be performed and must be =< upper limit of normal
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) or alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) =< 2.5 X ULN unless liver metastases are present, in which case it must be =< 5 x ULN (=< 14 days prior to registration)
* Calculated creatinine clearance of > 30 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) (=< 14 days prior to registration)
* Negative pregnancy test done =< 7 days prior to registration, for women of childbearing potential only

  * NOTE: The following restrictions apply while the patient is receiving study treatment and for the specified times before and after:

    * Female patient of child-bearing potential

      * Female patients of childbearing potential who are not abstinent and intend to be sexually active with a non sterilized male partner must use at least 1 highly effective method of contraception from the time of screening throughout the total duration of the drug treatment and the drug washout period (180 days after the last dose of study treatment). Non-sterilized male partners of a female patient of childbearing potential must use male condom plus spermicide throughout this period. Cessation of birth control after this point should be discussed with a responsible physician. Periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control. Female patients should also refrain from breastfeeding throughout this period
    * Male patients with a female partner of childbearing potential

      * Non-sterilized male patients who are not abstinent and intend to be sexually active with a female partner of childbearing potential must use a male condom plus spermicide from the time of screening throughout the total duration of the drug treatment and the drug washout period (180 days after the last dose of study treatment). However, periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of contraception. Male patients should refrain from sperm donation throughout this period
    * Female partners (of childbearing potential) of male patients must also use a highly effective method of contraception throughout this period
    * Females of childbearing potential are defined as those who are not surgically sterile (i.e., bilateral salpingectomy, bilateral oophorectomy, or complete hysterectomy) or post-menopausal
    * Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

      * Women < 50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution
      * Women >= 50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses > 1 year ago, had chemotherapy-induced menopause with last menses > 1 year ago
    * Highly effective methods of contraception, defined as one that results in a low failure rate (i.e., less than 1% per year) when used consistently and correctly are described below. Note that some contraception methods are not considered highly effective (e.g. male or female condom with or without spermicide; female cap, diaphragm, or sponge with or without spermicide; non-copper containing intrauterine device; progestogen-only oral hormonal contraceptive pills where inhibition of ovulation is not the primary mode of action [excluding Cerazette/desogestrel which is considered highly effective]; and triphasic combined oral contraceptive pills)
    * Effective methods include:

      * Copper T intrauterine device
      * Levonorgestrel-releasing intrauterine system (e.g., Mirena)
      * Implants: Etonogestrel-releasing implants: e.g. Implanon or Norplant
      * Intravaginal: Ethinylestradiol/etonogestrel-releasing intravaginal devices: e.g. NuvaRing
      * Injection: Medroxyprogesterone injection: e.g. Depo-Provera
      * Combined pill: Normal and low dose combined oral contraceptive pill
      * Patch: Norelgestromin/ethinylestradiol-releasing transdermal system: e.g. Ortho Evra
      * Minipill: Progesterone based oral contraceptive pill using desogestrel: Cerazette is currently the only highly effective progesterone-based
      * Tubal ligation
* Provide informed written consent
* Willing to return to enrolling institution for follow-up
* Willing to provide tissue, blood, and bone marrow samples for mandatory correlative research purposes

Exclusion Criteria:

* Any of the following uncontrolled intercurrent illness:

  * Clinically significant cardiovascular disease such as:

    * Symptomatic arrhythmias
    * Congestive heart failure
    * Myocardial infarction =< 3 months prior to registration
    * Any class 3 or 4 cardiac disease as defined by the New York Heart Association functional classification
    * Uncontrolled hypertension
    * Unstable angina pectoris

      * Note: Subjects with controlled, asymptomatic atrial fibrillation can enroll on study
  * Serious chronic gastrointestinal conditions associated with diarrhea
  * History of or ongoing confirmed progressive multifocal leukoencephalopathy (PML)
  * History of stroke or intracranial hemorrhage within 6 months before first dose of study drug
  * History of bleeding diathesis (e.g., hemophilia, von Willebrand disease)
  * Active uncontrolled infection (e.g., bacterial, viral or fungal, including subjects with positive cytomegalovirus [CMV] deoxyribonucleic acid [DNA] polymerase chain reaction [PCR]) requiring systemic therapy. NOTE: When the infection is controlled with systemic therapy, patients are permitted for this study
  * Active tuberculosis infection (clinical evaluation that includes clinical history, physical examination and radiographic findings, and tuberculosis [TB] testing in line with local practice)
  * Known human immunodeficiency virus (HIV/acquired immunodeficiency syndrome [AIDS]) infection as further severe immunosuppression with this regimen may occur
  * Hepatitis B or C serologic status:

    * Hepatitis B surface antigen and hepatitis B PCR positive will be excluded
    * Hepatitis B core antibody (anti-HBc) positive and who are surface antigen negative, and hepatitis B PCR positive will be excluded
    * These above patients once treated for hepatitis B and became hepatitis B PCR negative, they will be eligible
    * Hepatitis C PCR positive will be excluded. Once treated and hepatitis C PCR negative will be eligible
    * NOTE: Once patients with active hepatitis treated with effective therapy and adequate disease control, they will be allowed for participation
* Any of the following because this study involves an investigational agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown

  * Pregnant women
  * Nursing women
  * Men and women of childbearing potential who are unwilling to employ highly effective method of contraception starting with the screening visit through 180 days after the last dose of trial treatment
* Treated with other active investigational agents (excluding venetoclax, acalabrutinib. or ibrutinib) =< 5 half -lives of the previous investigational agents, please consult study chair for the specific investigational agent
* Prior durvalumab treatment. Note: If patients were treated with other prior PD1 blockade or PDL1 blockade, they will still be eligible
* Active or recent (=< 2 months) documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc.]) not being controlled. Exceptions:

  * Patients with vitiligo or alopecia
  * Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
  * Any chronic skin condition that does not require systemic therapy
  * Patients without active disease in the last 3 years may be included but only after consultation with the study physician
  * Patients with celiac disease controlled by diet alone
* Evidence of interstitial lung disease or active, non-infectious pneumonitis
* Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Active central nervous system (CNS) lymphoma or cerebrospinal fluid involvement with malignant lymphoma cells that requires therapy
* Clinically significant coagulopathy per investigator's assessment (stable anticoagulation except warfarin or other vitamin K antagonist will be allowed)
* Received an allogenic stem cell transplant within the last 2 years; Or prior history of allogeneic stem cell transplant with history of graft versus host disease (GVHD)
* Active chronic GVHD requiring treatment
* Chronically taking a strong CYP3A inhibitor or inducer and moderate inducer and cannot be switched to an alternative agent at least 4 days prior to trial therapy initiation that in the opinion of investigator/treating physicians precludes utilization of trial therapy
* Patients taking proton pump inhibitor will be excluded. NOTE: Patient may be switch to an H2 blocker or antiacid
* History of another primary malignancy except for:

  * Malignancy treated with curative intent and with no known active disease >= 5 years before the first dose of study drug and of low potential risk for recurrence
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
  * Adequately treated carcinoma in situ without evidence of disease
  * Indolent malignancy with expected life expectancy more than 2 years
* Current or prior use of immunosuppressive medication =< 5 half-lives of previous immunosuppressive medication. Note: Immunosuppressive medication is in reference to treatment of autoimmune or inflammatory disorders (e.g., with cyclosporine, tacrolimus, methotrexate, azathioprine) due to the potential suppressive effect on T-cells. Prior treatments administered as CLL- or lymphoma-directed treatment are not considered immunosuppressive medication under this criterion, as clarified below. The following are exceptions to this criterion:

  * Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
  * Systemic corticosteroids at physiologic doses not to exceed =< 30 mg/day of prednisone or its equivalent
  * Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
  * Receipt of live attenuated vaccine =< 30 days prior to registration. Note: Patients, if enrolled, should not receive live vaccine whilst receiving investigational product (IP) and up to 30 days after the last dose of IP
  * Received monoclonal antibody therapy for CLL or lymphoma > 7 days prior to registration
  * Received a chimeric antigen receptor T-cell therapy for CLL or lymphoma > 30 days prior to registration
  * Received bi-specific antibody therapy for CLL or lymphoma > 7 days prior to registration
  * Consult with the study chair if other specific medication in question
* Any radiation therapy =< 1 week prior to registration
* Any major surgery =< 28 days prior to registration (Note: Routine tissue or nodal biopsy or small procedures typically heal fast will not be counted as surgery)
* Body weight =< 30 kg
* Life expectancy < 12 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2023-01-05 (Actual); Primary Completion 2027-02-22 (Estimated); Study Completion 2027-02-22 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | At 6 months (end of cycle 6). Each cycle is 28 days.
  Progression will be defined by Lugano positron emission tomography (PET)-computed tomography (CT) based criteria or chronic lymphocytic leukemia (CLL) criteria. The proportion of successes will be estimated by the number of successes divided by the total number of evaluable patients. Ninety-five percent confidence intervals for the true success proportion will be calculated according to the approach of Duffy and Santner. If patients are censored prior to 6 months, a Kaplan Meier estimate for progression-free survival at 6 months along with the 95% confidence intervals will be reported.

SECONDARY OUTCOMES:
Overall response rate | Up to 1 year
  Overall response rate (for both Richter transformation [RT] and CLL, calculated separately) will be estimated by the total number of patients who achieve a complete metabolic response (CMR)/partial metabolic response (PMR) or complete response (CR)/complete response with incomplete marrow recovery (CRi)/nodular partial response (nPR)/partial remission (PR) divided by the total number of evaluable patients. Exact binomial 95% confidence intervals for the true overall response rate will be calculated. The PR rate and CR rate will also be estimated.
Overall survival | From registration to death due to any cause, assessed up to 5 years
  The distribution of overall survival will be estimated using the method of Kaplan-Meier.
Progression-free survival (PFS) | From registration to progression or death due to any cause, assessed up to 2 years
  The distribution of progression-free survival will be estimated using the method of Kaplan-Meier. PFS estimates will be calculated at 3, 6, 12, and 24 months.
Treatment-free survival | From registration to subsequent treatment or death due to any cause, assessed up to 5 years
  The distribution of treatment-free survival will be estimated using the method of Kaplan-Meier.
Incidence of adverse events | Up to 30 days after last dose of study drug
  All eligible patients that have initiated treatment will be considered evaluable for assessing adverse event (AE) rate(s). Platelets and hemoglobin will be graded according to the Grading Scale for Hematologic Adverse Events in CLL Studies. The maximum grade for each type of AE will be recorded for each patient, and frequency tables will be reviewed to determine patterns. Additionally, the relationship of the AE(s) to the study treatment will be taken into consideration.

CONTACTS AND LOCATIONS:
Overall Officials: Paul J. Hampel, MD, Principal Investigator — Mayo Clinic in Rochester
Locations (3):
- United States (3):
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials